CLINICAL TRIAL: NCT04631913
Title: Oats and Oat-fiber for Diabetes Prevention and Management: A Systematic Review and Meta-analysis of Randomized Controlled Trials
Brief Title: Meta-analysis of Oats for Diabetes Prevention and Management
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Toronto (Other)
Collaborators: Quaker Oats Company (Industry)
Responsible Party: Principal Investigator, John Sievenpiper, Associate Professor, University of Toronto
Other Study IDs: QUAKER - Oats & glycemia
Record Dates: First submitted 2020-11-16; First posted 2020-11-17 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Healthy; Diabetes; Metabolic Syndrome; Overweight and Obesity
Keywords: oats; viscous dietary fiber; beta-glucan; glycemic control; diabetes
MeSH Terms: conditions — Diabetes Mellitus; Metabolic Syndrome; Overweight; Obesity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Oats are a commonly consumed source of viscous soluble fibre, which has an established role in cardiovascular disease risk management including in cholesterol and glycemic control. Oat beta-glucan is recognized for its cholesterol-lowering effects with approved health claims in Canada, US and Europe. However, the efficacy of oat beta-glucan on glycemic control is not clear. We propose to conduct a systematic review and meta-analysis to explore the efficacy of whole grain oats and oat beta-glucan on markers of glycemic control in people with, without or at risk for diabetes.

DETAILED DESCRIPTION:
RATIONALE Although oat beta-glucan has approved health claims in Canada, US, and Europe [1-3] and is recognized by major cardiovascular guidelines [4,5] for its cholesterol-lowering, there are no approved health claims for the maintenance or achievement of normal blood glucose [6] and its role in the prevention and management of diabetes are less clear. We are not aware of any systematic reviews and meta-analyses of prospective cohort studies of the relation of the intake of whole oats, oat products, or oat beta-glucan with diabetes risk. Although there are several systematic reviews and meta-analyses of randomized trials showing that oats and oat beta-glucan improve markers of glycemic control and insulin resistance [7-9], the census for theses analyses do not include new RCTs [10]. Similar to an evidence synthesis that we conducted for all viscous fibers (inclusive of oat beta-glucan) [11], we propose to conduct the "gold-standard: in evidence synthesis (a systematic review and meta-analysis of randomized trials using Grading of Recommendations Assessment Development and Evaluation [GRADE] system) to quantify and assess the certainty of the evidence for the effect of oats and oat beta-glucan on established targets for glycemic control including HbA1c, fasting glucose, fasting insulin, and measures of insulin sensitivity in participants stratified by their risk of diabetes.

OBJECTIVES To quantify and assess the certainty of the evidence for the effect of oats and oat beta-glucan on established targets for glycemic control including HbA1c, fasting plasma glucose (FPG), 2h-plasma glucose (2h-PG), fasting plasma insulin, and measures of insulin sensitivity and beta-cell function in participants who have diabetes, are at risk of diabetes (prediabetes, metabolic syndrome, or overweight/obese), or are otherwise healthy.

DESIGN We will follow the Cochrane Handbook for Systematic Reviews of Interventions [12] and report according to the Preferred Reporting Items for Systematic Reviews and Meta-Analyses (PRISMA) [13]. The protocol will be registered at www.clinicaltrials.gov.

DATA SOURCES MEDLINE, EMBASE, and The Cochrane Central Register of Controlled Trials will be searched for eligible trials. We will also supplement our search with manual searches.

STUDY SELECTION We will include randomized controlled trials of ≥2-weeks assessing the effect of whole grain oats or oat beta-glucan compared with a suitable non-oat control on established targets for glycemic control including HbA1c, fasting plasma glucose, 2h-plasma glucose (2h-PG), fasting plasma insulin, and measures of insulin resistance in participants with or without diabetes.

DATA EXTRACTION Two or more investigators will independently extract relevant data. Authors will be contacted for additional information and any missing data will be computed/imputed using standard formulae [12].

RISK OF BIAS Two or more investigators will independently assess risk of bias using the Cochrane Risk of Bias 2.0 Tool.

OUTCOMES The outcomes will include established targets for glycemic control including HbA1c, fasting plasma glucose (FPG), 2h-plasma glucose (2h-PG), fasting plasma insulin, and measures of hepatic insulin sensitivity (HOMA-IR, hyperinsulinemic euglycemic clamp) whole body insulin sensitivity (Matsuda OGTT-ISI, frequently sampled intravenous glucose tolerance test [FSIGTT], hyperinsulinemic-euglycemic clamp) and beta-cell function (insulin secretion index, ISSI-2).

DATA SYNTHESIS Data will be pooled using the Generic Inverse Variance method stratified by risk of diabetes. Random effects models will be used with paired analyses applied to crossover designs [14]. Heterogeneity will be assessed (Cochran Q statistic) and quantified (I2 statistic). Sources of heterogeneity will be explored by sensitivity analyses. If ≥10 trial comparisons are available, a priori subgroup analyses will also be conducted to explore sources of heterogeneity (dose, comparator, intervention form (whole grain oat or oat beta-glucan) follow-up, baseline levels, design, body weight change, saturated fat intake, carbohydrate intake, protein intake, intervention food matrix, oat beta-glucan molecular weight and risk of bias). Meta-regression will assess the significance of subgroup analyses. Linear and nonlinear dose-response analyses will be assessed by generalized least squares trend (GLST) estimation models and spline curve modelling (MKSPLINE procedure), respectively. When ≥10 trial comparisons are available, publication bias will be assessed by inspection of funnel plots and the Egger and Begg tests. Adjustment for evidence of funnel plot asymmetry or small study effects will be conducted by the Duval and Tweedie trim-and-fill method.

GRADE ASSESSMENT To assess the certainty of the evidence, we will use the GRADE system, an evidence-based grading system adopted by >100 organizations (http://www.gradeworkinggroup.org/). It grades the evidence as high, moderate, low or very low quality based on the study design and a series of downgrades (risk of bias, imprecision, inconsistency, indirectness, publication bias) and upgrades (large magnitude of the effect, dose-response gradient, and attenuation by confounding). We will follow the GRADE handbook (https://gdt.gradepro.org/app/handbook/handbook.html) and use the GRADEpro (GRADEprofiler) software Version 3.2.

KNOWLEDGE TRANSLATION PLAN FOR IMPACT We will follow the Ottawa model of Research for knowledge translation [15]. The results will be disseminated through interactive presentations at local, national, and international scientific meetings and publication in high impact journals. Target audiences will include public health and clinical communities with an interest in nutrition and cardiovascular disease. Feedback will be incorporated and used to improve public health messages and key areas for future research will be defined. The PIs will network among opinion leaders to increase awareness and participate directly in the development of future guidelines.

SIGNIFICANCE The proposed project will aid in knowledge translation related to the role of whole grain oats and oat fiber as add-on therapy in the primary and secondary prevention of cardiovascular disease, strengthening the evidence-base for guidelines development in the U.S., Canada, Europe, and beyond and improving health outcomes, by educating healthcare providers and patients, stimulating industry innovation, and guiding future research design.

REFERENCES

1. Food Directorate Health Products and Food Branch, Health Canada Oat products and blood cholesterol lowering Bureau of Nutritional Sciences, Ottawa (2010). Available at https://www.canada.ca/en/health-canada/services/food-nutrition/food-labelling/health-claims/assessments/products-blood-cholesterol-lowering-summary-assessment-health-claim-about-products-blood-cholesterol-lowering.html
2. U.S. Food & Drug Administration, Health and Human Services. Food Labeling: Health Claims; Soluble Dietary Fiber From Certain Foods and Coronary Heart Disease. 21 CFR Part 101 [Docket No. 01Q-0313]. Available at https://www.gpo.gov/fdsys/pkg/FR-2002-10-02/pdf/02-25067.pdf
3. EFSA Panel on Dietetic Products, Nutrition and Allergies (NDA) Scientific Opinion on the substantiation of a health claim related to oat beta-glucan and lowering blood cholesterol and reduced risk of (coronary) heart disease pursuant to Article 14 of Regulation (EC) No 1924/2006 EFSA J, 8 (12) (2010), p. 1885, 10.2903/j.efsa.2010.1885 Available at www.efsa.europa.eu/efsajournal.htm
4. Anderson TJ, Grégoire J, Pearson GJ, Barry AR, Couture P, Dawes M, Francis GA, Genest J Jr, Grover S, Gupta M, Hegele RA, Lau DC, Leiter LA, Lonn E, Mancini GB, McPherson R, Ngui D, Poirier P, Sievenpiper JL, Stone JA, Thanassoulis G, Ward R. 2016 Canadian Cardiovascular Society Guidelines for the Management of Dyslipidemia for the Prevention of Cardiovascular Disease in the Adult. Can J Cardiol. 2016 Nov;32(11):1263-1282
5. Catapano AL, Graham I, De Backer G, Wiklund O, Chapman MJ, Drexel H, Hoes AW, Jennings CS, Landmesser U, Pedersen TR, Reiner Ž, Riccardi G, Taskinen MR, Tokgozoglu L, Verschuren WMM, Vlachopoulos C, Wood DA, Zamorano JL, Cooney MT; ESC Scientific Document Group. 2016 ESC/EAS Guidelines for the Management of Dyslipidaemias. Eur Heart J. 2016 Oct 14;37(39):2999-3058
6. European Food Safety Authority (EFSA). Scientiﬁc Opinion on the Substantiation of Health Claims Related to Beta-Glucans and Maintenance or Achievement of Normal Blood Glucose Concentrations (ID 756, 802, 2935) Pursuant to Article 13(1) of Regulation (EC) No 1924/2006.2010; European Food Safety Authority (EFSA): Parma, Italy, 2010
7. Hou Q1, Li Y2, Li L3, Cheng G4, Sun X5, Li S6, Tian H7. The Metabolic Effects of Oats Intake in Patients with Type 2 Diabetes: A Systematic Review and Meta-Analysis. Nutrients. 2015 Dec 10;7(12):10369-87. doi: 10.3390/nu7125536
8. Shen XL, Zhao T, Zhou Y, Shi X, Zou Y, Zhao G. Effect of Oat β-Glucan Intake on Glycaemic Control and Insulin Sensitivity of Diabetic Patients: A Meta-Analysis of Randomized Controlled Trials. Nutrients. 2016 Jan 13;8(1). pii: E39. doi: 10.3390/nu8010039. Review
9. He LX, Zhao J, Huang YS, Li Y. The difference between oats and beta-glucan extract intake in the management of HbA1c, fasting glucose and insulin sensitivity: a meta-analysis of randomized controlled trials. Food Funct. 2016 Mar;7(3):1413-28. doi: 10.1039/c5fo01364j.
10. Li X, Cai X, Ma X, Jing L, Gu J, Bao L, Li J, Xu M, Zhang Z, Li Y. Short- and Long-Term Effects of Wholegrain Oat Intake on Weight Management and Glucolipid Metabolism in Overweight Type-2 Diabetics: A Randomized Control Trial. Nutrients. 2016 Sep 7;8(9):pii:E549
11. Jovanovski E, Khayyat R, Zurbau A, Komishon A, Mazhar N, Sievenpiper JL, Blanco Mejia S, Ho HVT, Li D, Jenkins AL, Duvnjak L, Vuksan V. Should Viscous Fiber Supplements Be Considered in Diabetes Control? Results From a Systematic Review and Meta-analysis of Randomized Controlled Trials. Diabetes Care. 2019 May;42(5):755-766
12. Higgins JPT, Greens S (editors). Cochrane Handbook for Systematic Reviews of Interventions Version 5.1.0 [updated March 2011]. The Cochrane Collaboration, 2011. Available from www.cochrane-handbook.org.
13. Moher D, Liberati A, Tetzlaff J, Altman DG; PRISMA Group. Preferred reporting items for systematic reviews and meta-analyses: the PRISMA statement. BMJ. 2009;339:b2535.
14. Elbourne DR, Altman DG, Higgins JP, Curtin F, Worthington HV, Vail A. Meta-analyses involving cross-over trials: Methodological issues. Int J Epidemiol. 2002;31:140-149.
15. Graham ID, Logan J. Innovations in knowledge transfer and continuity of care. Can J Nurs Res. 2004;36(2):89-103.

ELIGIBILITY:
Inclusion Criteria:

* Oat or oat beta-glucan intervention
* Adult human dietary trial
* Randomized treatment allocation
* ≥ 2 weeks intervention period
* Suitable control (i.e. non-oat control)
* Viable endpoint data

Exclusion Criteria:

* Non-human studies
* Non-randomized treatment allocation
* < 2 weeks intervention period
* Lack of a suitable control
* No viable endpoint data

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult humans with, without or at risk fo diabetes
Sampling Method: Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2020-08-14 (Actual); Primary Completion 2021-07-31 (Estimated); Study Completion 2021-11-30 (Estimated)

PRIMARY OUTCOMES:
Glycemic control - HbA1c | At least 2 weeks
  Mean difference
Glycemic control - Fasting plasma glucose | At least 2 weeks
  Mean difference
Glycemic control - 2h-plasma glucose (2h-PG) | at least 2 weeks
  Mean difference
Glycemic control - Fasting blood insulin | At least 2 weeks
  Mean difference
Insulin Sensitivity - hepatic | At least 2 weeks
  Ratio of means (aggregate of HOMA-IR, hyperinsulinemic euglycemic clamp hepatic insulin sensitivity)
Insulin Sensitivity - whole body | At least 2 weeks
  Ratio of means (aggregate of Matsuda OGTT-ISI, frequently sampled intravenous glucose tolerance test (FSIGTT), hyperinsulinemic euglycemic clamp hyperinsulinemic clamp whole body insulin sensitivity)
Beta-cell function | At least 2 weeks
  Ratio of means (aggregate of insulin secretion index, ISSI2)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Toronto, Toronto, Ontario, Canada